CLINICAL TRIAL: NCT01752114
Title: Early Diagnosis of Pulmonary Nodules Using A Plasma Proteomic Classifier, Protocol Number 1001-12
Brief Title: Early Diagnosis of Pulmonary Nodules
Status: Completed | Type: Observational
Sponsor: Integrated Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: PANOPTIC (1001-12)
Record Dates: First submitted 2012-11-30; First posted 2012-12-19 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2016-08

CONDITIONS: Precancerous Conditions; Carcinoma
Keywords: Precancerous conditions; Carcinoma
MeSH Terms: conditions — Precancerous Conditions; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is intended to determine the positive predictive value (PPV) and negative predictive value (NPV) of the multiprotein classifier based on the observed study prevalence of Non-Small Cell Lung Cancer (NSCLC) in the study participants.

DETAILED DESCRIPTION:
Patients must present with previously non-diagnosed lung nodules as found on CT. There is no change to the typical standard of care that any of the investigating physicians and/or centers provide the patients enrolled in this study. The data from this study will not be used to diagnose cancer nor be used to influence treatment decisions for the study participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Smoking history: Never, Former, Current
* Subject undergoing diagnostic evaluation for a lung nodule
* Subject undergoing evaluation for a lung nodule by a pulmonologist, and/or by a thoracic surgeon
* Baseline CT scan identifying lung nodule performed within 60 days of subject enrollment
* Nodule(s) identified by CT scan previously not followed
* Subject willing to provide informed consent for the collection of blood specimens

Exclusion Criteria:

* Nodule work-up at the time of enrollment eligibility indicates any prior attempted or completed diagnostic biopsy procedure, such as transthoracic needle aspiration, bronchoscopic biopsy or surgery
* A prior CT scan is available that previously identifies the same lung nodule under consideration for study inclusion on the most current CT scan; AND the prior CT scan was performed more than 60 days before the current CT scan, irrespective of the candidate nodule's radiographic characterization such as size, density or appearance
* Current diagnosis of any cancer
* Prior diagnosis of any cancer within 2 years of lung nodule detection, except for non-melanoma skin cancer
* Administration of blood products, e.g. packed red blood cells, fresh frozen plasma, or platelets, within 30 days of subject enrollment
* History of human immunodeficiency virus (HIV) or Hepatitis C

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject undergoing evaluation for a lung nodule by a pulmonologist in a pulmonary or chest clinic, and/or by a thoracic surgeon at the time of enrollment
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2012-10; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of adult patients diagnosed with Non-Small Cell Lung Cancer | 2 years post enrollment
  Incidence rate of Non-Small Cell Lung Cancer as determined by histologic or cytologic diagnosis and/or radiographically stability at 2 years post enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Russell F. Hudnall, Study Director — Integrated Diagnostics, Inc.
Locations (33):
- United States (31):
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Pulmonary Associates of Southern Arizona, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Georgia Lung Associates, Austell, Georgia
  - Suburban Lung Associates, Elk Grove Village, Illinois
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Pulmonary & Crit Care Associates of Baltimore, Baltimore, Maryland
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Baystate Health, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Beaumont Health System, Royal Oak, Michigan
  - Virginia Piper Cancer Institute - Allina Health, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Medical Center, Chesterfield, Missouri
  - New York University Clinical Cancer Center, New York, New York
  - Charleston Research Institute, Charleston, North Carolina
  - Carolinas HealthCare System, Charlotte, North Carolina
  - LeBaurer Healthcare, Greensboro, North Carolina
  - Salem Chest Specialists, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Clinic, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Scott & White Clinic, Temple, Texas
  - Inova Healthcare, Fairfax, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Canada (2):
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Institute Universitarie de Cardiologie et de Pneumologie, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Long KJ, Silvestri GA, Kammer MN, Gibbs S, Wu W, Johal M, Pipavath S, Pitcher T, Jett J, Nair VS. Validation of a High-Specificity Blood Autoantibody Test to Detect Lung Cancer in Pulmonary Nodules. CHEST Pulm. 2025 Mar;3(1):100130. doi: 10.1016/j.chpulm.2024.100130. Epub 2024 Dec 25. PMID 40296864
- [Derived] Silvestri GA, Tanner NT, Kearney P, Vachani A, Massion PP, Porter A, Springmeyer SC, Fang KC, Midthun D, Mazzone PJ; PANOPTIC Trial Team. Assessment of Plasma Proteomics Biomarker's Ability to Distinguish Benign From Malignant Lung Nodules: Results of the PANOPTIC (Pulmonary Nodule Plasma Proteomic Classifier) Trial. Chest. 2018 Sep;154(3):491-500. doi: 10.1016/j.chest.2018.02.012. Epub 2018 Mar 1. PMID 29496499